CLINICAL TRIAL: NCT00566111
Title: Modulation of Glutamatergic Neurotransmission in the Treatment of Bipolar Depression
Brief Title: Ceftriaxone in the Management of Bipolar Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early indication of an unfavorable risk/benefit ratio.
Sponsor: Yale University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0704002567
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2016-08

CONDITIONS: Bipolar Depression
Keywords: Ceftriaxone; Acute Antidepressant Effects; Glutamatergic System; Double-Blind; Mood Disorders; Bipolar Disorder; Depression; Affective Disorders
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Depression | interventions — Ceftriaxone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: ceftriaxone
- P (Placebo Comparator)
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: ceftriaxone — 2g per day which will be administered IV via midline, 7 days a week for 4 weeks.
  Other Names: Rocephin; Ceftriaxone Sodium
  Arms: A
Drug: Saline solution — Saline solution will be administered IV via midline, 7 days a week for 4 weeks.
  Arms: P

SUMMARY:
We aim to study the efficacy of intravenous ceftriaxone in a four-week, inpatient, placebo-controlled, double-blind study, as an augmentation therapy in patients with bipolar disorder, currently depressed, who have failed to respond to conventional treatments.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of bipolar disorder
* Presence of a current major depressive episode on the SCID
* Score of 17 or greater on the HDRS
* Failure to respond to two previous medication trials
* Capable of giving voluntary written consent

Exclusion Criteria:

* Hypersensitivity to penicillin or cephalosporin, resulting in anaphylaxis
* Significant current substance dependence/abuse within 3 months preceding the trial
* Significant history of intravenous drug abuse
* Active suicidal ideation
* Pregnant/lactating mothers
* Significant medical history
* Patients on anticoagulation treatment
* Patients who test positive for HIV or Hep B or C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zubin Bhagwagar, MD PhD, Principal Investigator — Yale University; Gerard Sanacora, MD PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Mineur YS, Picciotto MR, Sanacora G. Antidepressant-like effects of ceftriaxone in male C57BL/6J mice. Biol Psychiatry. 2007 Jan 15;61(2):250-2. doi: 10.1016/j.biopsych.2006.04.037. Epub 2006 Jul 24. PMID 16860779
- [Background] Rothstein JD, Patel S, Regan MR, Haenggeli C, Huang YH, Bergles DE, Jin L, Dykes Hoberg M, Vidensky S, Chung DS, Toan SV, Bruijn LI, Su ZZ, Gupta P, Fisher PB. Beta-lactam antibiotics offer neuroprotection by increasing glutamate transporter expression. Nature. 2005 Jan 6;433(7021):73-7. doi: 10.1038/nature03180. PMID 15635412

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Saline solution: Saline solution will be administered IV via midline, 7 days a week for 4 weeks.
Period: Overall Study
Arm/Group | Ceftriaxone | Placebo
Started | 2 | 3
Completed | 2 | 1
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftriaxone | Placebo | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale (HDRS) Score From Baseline.
Description: Number of patients with scores that decreased at four weeks.
Time Frame: 4 weeks
Population: only participants with complete data at 4 weeks were analyzed
Measure: Number; unit: participants
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 2 | 1
participants | 2 | 1

2. Secondary Outcome: Change in Score on the 16-item Quick Inventory of Depressive Symptoms (QIDS) From Baseline.
Description: Number of patients with scores that decreased at four weeks.
Time Frame: 4 weeks
Population: These data were not collected.
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Subjects Who Achieve Remission as Defined by a HDRS Score < 7.
Time Frame: 4 weeks
Population: only participants with complete data at 4 weeks were analyzed
Measure: Number; unit: participants
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 2 | 1
participants | 0 | 0

4. Secondary Outcome: Change in Montgomery Asberg Depression Rating Scale (MADRS)Score From Baseline.
Description: The number of patients that had a decrease on MADRS at 4 weeks.
Time Frame: 4 weeks
Population: only participants with complete data at 4 weeks were analyzed
Measure: Number; unit: participants
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 2 | 1
participants | 2 | 0

5. Secondary Outcome: Change in Ratings on the Clinical Global Impressions Scale for Bipolar Disorder (CGI-BP).
Description: The number of patients that had a decrease on CGI-BP at 4 weeks.
Time Frame: 4 weeks
Population: only patients with complete data at 4 weeks were analyzed
Measure: Number; unit: participants
Arm/Group | Ceftriaxone | Placebo
Number analyzed (Participants) | 2 | 1
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 4 weeks.
Arm/Group | Ceftriaxone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftriaxone (N=2) | Placebo (N=3)
Drowsiness (General disorders) | 1 (1) | 1 (1)
Difficulty Concentrating (General disorders) | 2 (2) | 2 (2)
Poor Coordination (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nightmares (Psychiatric disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
Tremors (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes